CLINICAL TRIAL: NCT01501760
Title: Effect of Bevacizumab Subconjunctival Injections on Corneal Newvessels
Brief Title: Efficacy and Safety Study of Avastin to Treat Neovascularisation of the Cornea
Acronym: BECONNEC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: I07034
Record Dates: First submitted 2011-12-26; First posted 2011-12-29 (Estimated); Last update posted 2019-10-24 (Actual); Status verified 2018-10

CONDITIONS: Corneal Newvessels
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- bevacizumab (Experimental): Three subconjunctival injections of 0.5 ml of bevacizumab at inclusion, 1 month, 2 month.
  Interventions: Drug: bevacizumab
- Placebo (Placebo Comparator): Three subconjunctival injections of 0.5 ml of Nacl at inclusion, 1 month, 2 month.
  Interventions: Drug: NaCl

INTERVENTIONS:
Drug: bevacizumab — Three subconjunctival injections of 0.5 ml of bevacizumab at: inclusion, 1 month, 2 month
  Arms: bevacizumab
Drug: NaCl — Three subconjunctival injections 0.5 ml placebo (Balanced salt) solution at inclusion, 1 month, 2month
  Arms: Placebo

SUMMARY:
Corneal newvessels may arise from a fan of pathologies, inducing long-standing corneal opacification requiring keratoplasty. These last years, VEGF inhibitors have been designed to reduce newascularization induced by gastric cancer or age-related macular degeneration. A few reports have been published showing the interest of VEGF inhibitors to treat corneal newvessels, but no randomized study has been achieved to date.

This study is designed to assess the efficacy of Bevacizumab, a VEGF inhibitor monoclonal antibody, to reduce the surface of corneal newvessels in when compared to placebo

DETAILED DESCRIPTION:
This study will involve 42 outpatients of the CHU of Limoges, Bordeaux, and Toulouse, addressed for corneal pathologies including corneal newvessels. The patients will be randomly assigned to two groups, one receiving three subconjunctival injections of bevacizumab, the other three subconjunctival injections of placebo (Balanced salt solution). The progression of newvessels will be assessed using color photographs and a picture-analyser software that will calculate the percentage of corneal surface occupied by the newvessels. Randomization, and preparation of both study drug and placebo syringes will be performed by the central pharmacy of the CHU de Limoges. Patients will be followed-up as outpatients, with visits scheduled 15 days before treatment, at baseline, and then at 1 month, 2 months, 3 months, and 6 months.

* Primary outcome: To demonstrate Bevacizumab subconjunctival injections effectiveness on corneal neovascularisation reduction definite by a superior percentage of patient with a reduction higher than 30 % of the corneal surface occupied by newvessels , at 3 months, in the group Bevacizumab compared with the group placebo
* Secondary outcomes:
* The effectiveness of bevacizumab on reducing the percentage of corneal surface occupied by neovascularization at 6 months
* The effectiveness of bevacizumab on reducing the use of corneal graft.
* The local and general toxicity of bevacizumab administered by subconjunctival way.

ELIGIBILITY:
Inclusion Criteria:

inclusion criteria:

* Patients with corneal neovascularization whatever the origin
* Patient did not receive treatment with topical corticosteroids during the month preceding inclusion.
* Patient who has been properly informed and signed consent
* Patient aged over 18
* Patient affiliated with a health insurance plan or benefit of such a regime

Exclusion Criteria:

* Patients who received local or general treatment of concomitant prostaglandin derivatives

  * Patients with current infection of the cornea or other tissue / organ
  * Women of childbearing age without contraception
  * Pregnancy and Lactation
  * Patient participating in another study
  * Patient with contact lenses
  * Patients with uncontrolled hypertension
  * Patient with a history of stroke, myocardial infarction, angina pectoris, thrombophlebitis, Raynaud's phenomenon.
  * Patients hypersensitive to the active substance or any excipients
  * Patients hypersensitive to products of Chinese hamster ovary cells or other recombinant human or humanized antibodies.
  * Patients with active bacterial eye infections, fungal, parasitic or viral infection (with the exception of herpes)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2012-05-13 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Neovascularisation reduction at 3 months | at 3 months
  Assessement using color photographs and a picture-analyser software that will calculate the percentage of corneal surface occupied by the newvessels at 3 months. A reduction of 30% is target.

SECONDARY OUTCOMES:
Local and general toxicity of bevacizumab | at 1 months, 2 month, 3 month, 6 month
  Safty data are collected at each visit either by clinical examination or by patient questionnary
Efficacy at 6 months | at 6 month
  Assessed using color photographs and a picture-analyser software that will calculate the percentage of corneal surface occupied by the newvessels at 6 month

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Service d'Ophtalmologie, Limoges
  - CHU Poitiers-Ophtalmologie, Poitiers
  - CHU St Etienne, Saint-Etienne
  - CHU Strasbourg- Service Ophtalmlogie, Strasbourg
  - CHU de Toulouse, Service d'Ophtalmologie, Toulouse